CLINICAL TRIAL: NCT06157996
Title: Tislelizumab Plus CapeOX ± Lenvatinib as First-Line Treatment for Advanced GC/GEJC With Positive PD-L1 and Low TMEscore: A Multi-center, Prospective, Phase II Study
Brief Title: Lenvatinib Plus Tislelizumab and CapeOX as First-Line Treatment for Advanced GC/GEJC With Positive PD-L1 and Low TMEscore
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-478
Record Dates: First submitted 2023-11-26; First posted 2023-12-06 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer
Keywords: Lenvatinib; Tislelizumab; First-line treatment; GC/GEJC; TME score; PD-L1 positive
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive treatment of lenvatinib and tislelizumab plus CapeOX chemotherapy (Experimental): Efficacy of lenvatinib and tislelizumab plus CapeOX as first-line treatment
  Interventions: Drug: lenvatinib and tislelizumab plus CapeOX chemotherapy
- Conventional treatment of tislelizumab plus CapeOX chemotherapy (Active Comparator): Efficacy of tislelizumab plus CapeOX as first-line treatment
  Interventions: Drug: tislelizumab plus CapeOX chemotherapy

INTERVENTIONS:
Drug: lenvatinib and tislelizumab plus CapeOX chemotherapy — Tislelizumab 200mg, iv, d1+ oxaliplatin 130mg/m2, iv, d1+ capecitabine 1000mg/m2, bid po, D1-14, q3w + Lenvatinib 8mg, qd po regimen are received, respectively (3 weeks as a cycle, a maximum of 8 cycles of treatment). Then the maintenance treatment phase with tislelizumab + lenvatinib is entered, and the specific dosage is the same as the treatment period.
  Arms: Intensive treatment of lenvatinib and tislelizumab plus CapeOX chemotherapy
Drug: tislelizumab plus CapeOX chemotherapy — Tislelizumab 200mg, iv, d1+ oxaliplatin 130mg/m2, iv, d1+ capecitabine 1000mg/m2, bid po, D1-14, q3w regimen are received, respectively (3 weeks as a cycle, a maximum of 8 cycles of treatment). Then the maintenance treatment phase with tislelizumab is entered, and the specific dosage is the same as the treatment period.
  Arms: Conventional treatment of tislelizumab plus CapeOX chemotherapy

SUMMARY:
This is a multicenter, prospective, phase II clinical study to evaluate the efficacy and safety of intensive treatment with lenvatinib plus tislelizumab and CapeOX as first-line treatment for advanced gastric cancer or gastroesophageal junction adenocarcinoma with PD-L1 positive and low TMEscore. A total of 92 subjects are randomly divided into study group and control group according to 1:1 ratio. Tislelizumab 200mg, iv, d1+ oxaliplatin 130mg/m2, iv, d1+ capecitabine 1000mg/m2, bid po, D1-14, q3w ± Lenvatinib 8mg, qd po regimen are received, respectively (3 weeks as a cycle, a maximum of 8 cycles of treatment). Then the maintenance treatment phase with tislelizumab ± lenvatinib is entered, and the specific dosage is the same as the treatment period. Effectiveness is assessed every 9 weeks (±7 days) until disease recurrence, metastasis, death, or loss of follow-up. The primary endpoint of this study was PFS, and secondary endpoints were OS, ORR, DoR, and DCR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study, signed the informed consent, and had good compliance;
2. Age over 18 (including 18 years old), gender is not limited;
3. Histologically and/or cytologically confirmed advanced gastric cancer or gastroesophageal junction adenocarcinoma (stage IV);
4. Tumor with PD-L1 positive and low tumor microenvironment score (TMEscore)
5. Have not received systemic antitumor therapy before; Or have previously received adjuvant or neoadjuvant therapy (chemotherapy/radiotherapy) for the purpose of cure, and the time of tumor recurrence > 6 months since the last treatment
6. ECOG performance status of 0-2 points;
7. Expected survival ≥12 weeks;
8. Blood test (without blood transfusion within 14 days) 1) Neutrophil absolute value ≥1.5×10^9/L, platelet ≥100×10^9/L, hemoglobin ≥90g/L); 2) Liver function test (aspartate aminotransferase and glutamate aminotransferase ≤3×ULN, bilirubin ≤1.5×ULN; In case of liver metastasis, AST and ALT≤5×ULN); 3) Renal function (serum creatinine ≤1.5×ULN, or creatinine clearance (CCr)≥60ml/min);
9. Men and women of childbearing age must use effective contraceptive methods.

Exclusion Criteria:

1. Previously received therapy that targets T cell co-stimulation or checkpoint pathways ,such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.;
2. Previously received anti-vascular small-molecule targeted drug therapy, such as fuquinitinib, regofenib, etc.;
3. Received major surgery within 4 weeks prior to the first drug administration; radiotherapy, radiofrequency ablation and other investigational drugs for tumors within 2 weeks;
4. Received live vaccine within 4 weeks prior to the first drug administration (except inactivated viral vaccine for seasonal influenza);
5. A history of severe intolerance to drugs involved in the study (i.e., grade 4 toxicity of one of these drugs; Class 3-4 toxicity of other co-administered drugs is not excluded);
6. Known allergy to the study drug or any of its excipients;
7. HER2 positive gastric cancer or gastroesophageal junction adenocarcinoma;
8. The patient had other malignancies within the previous 5 years or at the same time (except cured basal cell carcinoma, stage I squamous cell carcinoma, in situ carcinoma, intramucosal carcinoma, and superficial bladder cancer);
9. Known brain or meningeal metastases;
10. Patients who are preparing for or have previously received an organ or bone marrow transplant;
11. A history of human immunodeficiency virus (HIV) infection;
12. A history of psychotropic substance abuse or drug use;
13. Condition that may interfere with the detection and management of suspected drug-related pulmonary toxicity, such as interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severe impairment of lung function;
14. Known active or suspected autoimmune disease (except for patients with stable disease at enrollment who do not require systemic immunosuppressive therapy);
15. Patients who required systemic corticosteroids (> 10 mg/ day efficacy dose of prednisone) or other immunosuppressive agents within 2 weeks prior to initial administration or during the study period. However, adrenal hormone replacement therapy with topical or inhaled steroids, or a therapeutic dose of prednisone ≤ 10mg/ day in the absence of active autoimmune disease was permitted;
16. Any active infection that requires systematic anti-infective treatment occurs within 2 weeks prior to the first dose (expect prophylactic antibiotic therapy, such as for urinary tract infections or chronic obstructive pulmonary disease);
17. Active heart disease, including myocardial infarction, severe/unstable angina in the 6 months prior to treatment. Echocardiography showed that the left ventricular ejection fraction was less than 50%, indicating poor arrhythmia control.
18. Obvious clinical bleeding symptoms or obvious bleeding tendency and hemoptysis within 3 months prior to treatment. Or treatment of venous/venous thrombosis events within the preceding 6 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; Long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day) is required;
19. Any other disease, a clinically significant metabolic abnormality, abnormal physical examination or abnormal laboratory examination, for which, in the investigator's judgment, there is reason to suspect that the patient has a disease or condition unsuitable for the use of the investigational agent;
20. Anything that, in the investigator's opinion, could put subjects receiving the study drug at risk, interfere with the study drug, subject safety assessment, or interpretation of the results;
21. Pregnant or lactating women or women who may become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 3 years
  Defined as the time between the onset of PD or death when a patient first receives the study drug, whichever occurs first

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Defined as the time between the patient's first receipt of the study drug to death
Objective Response Rate (ORR) | 3 years
  Defined as the proportion of patients who achieved complete response (CR) or partial response (PR)
Disease Control Rate (DCR) | 3 years
  Defined as the proportion of patients achieving CR, PR, or stable disease (SD).
Duration of response (DoR) | 3 years
  Defined as the time between when a patient first reaches CR or PR to PD

CONTACTS AND LOCATIONS:
Overall Officials: Wangjun Liao, MD, PhD, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No